CLINICAL TRIAL: NCT06730243
Title: To Evaluate the Impact of Retzius-sparing Robot-assisted Radical Prostatectomy With "Sandwich" Technique of Total Urethral Reconstruction on Early Recovery of Urinary Continence (UC) Compared to the Conventional Approach (Anterior Approach) and Laparoscopic Radical Prostatectomy for the Treatment of Clinically Localized Prostate Cancer (PCa).
Brief Title: Retzius-sparing Robot-assisted Radical Prostatectomy With "Sandwich" Technique of Total Urethral Reconstruction Versus Standard Robot-Assisted Radical Prostatectomy Versus Laparoscopic Radical Prostatectomy Surgery: A Comparative Prospective Study of 300 Patients
Acronym: RS-RARP-S
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Xing Nianzeng, National Cancer Center, Ministry of Science and Technology of the People´s Republic of China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24/048-4328
Record Dates: First submitted 2024-12-08; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Retzius-sparing Robot-assisted Radical Prostatectomy With "Sandwich" Technique of Total Urethral Reconstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RS-RARP-S (Experimental): Retzius-sparing robot-assisted radical prostatectomy and "Sandwich" Technique of Total Urethral Reconstruction
  Interventions: Procedure: Retzius-sparing robot-assisted radical prostatectomy and "Sandwich" Technique of Total Urethral Reconstruction
- S-RARP (Experimental): Standard RARP
  Interventions: Procedure: Standard Robot-Assisted Radical Prostatectomy
- LRP (Sham Comparator): Laparoscopic Radical Prostatectomy
  Interventions: Procedure: Laparoscopic Radical Prostatectomy

INTERVENTIONS:
Procedure: Retzius-sparing robot-assisted radical prostatectomy and "Sandwich" Technique of Total Urethral Reconstruction — Retzius-sparing robot-assisted radical prostatectomy and "Sandwich" Technique of Total Urethral Reconstruction
  Arms: RS-RARP-S
Procedure: Standard Robot-Assisted Radical Prostatectomy — Standard Robot-Assisted Radical Prostatectomy
  Arms: S-RARP
Procedure: Laparoscopic Radical Prostatectomy — Laparoscopic Radical Prostatectomy
  Arms: LRP

SUMMARY:
To evaluate the impact of Retzius-sparing robot-assisted radical prostatectomy with "Sandwich" Technique of Total Urethral Reconstruction on early recovery of urinary continence (UC) compared to the conventional approach (anterior approach) and Laparoscopic Radical Prostatectomy for the treatment of clinically localized prostate cancer (PCa).Purpose: The trial compares outcomes between three groups.

DETAILED DESCRIPTION:
300 consecutive patients with clinically localized PCa underwent RS-RARP-S (Retzius-sparing robot-assisted radical prostatectomy and "Sandwich" Technique of Total Urethral Reconstruction) or S-RARP (Standard RARP) or LRP by 6 experienced surgeons regardless of clinicopathological features. The indication for one technique or the others were surgeon preference; one surgeon exclusively performed RS-RARP-S( did not exclude high risk cases or those with apical and anterior tumors), two surgeons performed S-RARP, and three surgeons exclusively performed LRP. The investigation include an extensive evaluation of clinical, oncological, functional and quality of life related data by means of validated patient-reported outcome measures.

The primary outcome is early recovery of urinary continence compared to the conventional approach.

ELIGIBILITY:
Inclusion Criteria:

* Histological verified prostate carcinoma (first diagnosis) Indication for primary curative radical prostatectomy Age ≤80 years Patient agrees to randomisation Patient is able to fill in the questionnaires on his own Patient is willing to provide written informed consent

Exclusion Criteria:

* Insufficient knowledge of German Severe cognitive impairment Obesity (BMI > 35) Current existing severe comorbidities (e.g. liver cirrhosis, second malignancy or relapse of every kind) Tumor stage: T4 Previous malignancy (≤ 3 years before trial participation) Neoadjuvant therapy (hormons) within the last 3 months before participation in the trial Patient is immuno-compromised History of intermittent urinary self-catheterization within the last year Psychological disorders (dementia, chronic depression, psychosis) Any of the following treatments ≤ 3 months before trial participation: surgery of the sigmoid colon, extended haemorrhoid resection, transurethral needle ablation of the prostate (TUNA), osteosynthesis of the pelvis, salvage prostatectomy Patients with chronic urinary infection Dialysis patients Lacking willingness for data storage and handling in the frame of the trial protocol/aims

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
immediate urinary continence analysis | 1day，1month, 3 months after removal of the urinary cathete
  Primary outcome was UC (defined as 0 pads/one security liner per day) after catheter removal

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided